CLINICAL TRIAL: NCT06502028
Title: Video Laryngeal Mask Versus Endotracheal Tube in Patients Undergoing Laparoscopic Cholecystectomy Surgery Under General Anesthesia: a Prospective Randomized Controlled Trial
Brief Title: Video Laryngeal Mask Versus Endotracheal Tube Undergoing Laparoscopic Cholecystectomy Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2308-160-1461
Record Dates: First submitted 2024-06-27; First posted 2024-07-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Cholecystitis
MeSH Terms: conditions — Cholecystitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Video LMA (Experimental): The airway is secured with a video laryngeal mask airway (VLMA).
  Interventions: Device: Video laryngeal mask airway
- Control (Active Comparator): The participant is intubated with an endotracheal tube via direct laryngoscopy.
  Interventions: Device: Endotracheal tube

INTERVENTIONS:
Device: Video laryngeal mask airway — The airway is secured with a video laryngeal mask airway.
  Arms: Video LMA
Device: Endotracheal tube — The participant is intubated with an endotracheal tube via direct laryngoscopy.
  Arms: Control

SUMMARY:
The aim of this study is to investigate the effectiveness of using a video laryngeal mask for airway management in patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
The investigators will compare the time required to secure the airway when inserting a video laryngeal mask (LMA) versus performing endotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 19 years old
* Patients planned for elective laparoscopic cholecystectomy

Exclusion Criteria:

* High risk of aspiration (e.g. gastro-esophageal reflux disease, hiatus hernia, pregnancy, history of gastrectomy)
* Difficult airway (e.g. limitation of mouth opening, limitation of neck extension, oropharyngeal pathology)
* Obesity (BMI > 30 kg/m2)
* Tooth mobility

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-12-26 (Estimated); Study Completion 2026-05-26 (Estimated)

PRIMARY OUTCOMES:
Time required for VLMA insertion or intubation | After induction of anesthesia, before the operation starts.
  Time required for VLMA insertion or intubation

SECONDARY OUTCOMES:
Number of trials | After induction of anesthesia, before the operation starts.
  Video laryngeal mask airway insertion or endotracheal intubation
Peak airway pressure | After video laryngeal mask airway insertion or intubation, before extubation
  Peak airway pressure
Minute ventilation | After video laryngeal mask airway insertion or intubation, before extubation
  Minute ventilation
End tidal carbon dioxide | After video laryngeal mask airway insertion or intubation, before extubation
  End tidal carbon dioxide
Oropharyngeal leak pressure | After video laryngeal mask airway insertion or intubation, before extubation
  Oropharyngeal leak pressure
Traces of blood on airway device after extubation | After extubation, before transfer to PACU
  Traces of blood on airway device after extubation
Postoperative sore throat | 1 hour after end of operation
  4-point scale, 0 = no sore throat; 1 = mild sore throat (complaints of sore throat only on asking); 2 = moderate sore throat (complaints of sore throat on his/her own); 3 = severe sore throat (change of voice or hoarseness, associated with throat pain)
Postoperative sore throat | 24 hours after end of operation
  4-point scale, 0 = no sore throat; 1 = mild sore throat (complaints of sore throat only on asking); 2 = moderate sore throat (complaints of sore throat on his/her own); 3 = severe sore throat (change of voice or hoarseness, associated with throat pain)
Postoperative hoarseness | 1 hour after end of operation
  4-point scale, 0 = no hoarseness; 1 = mild hoarseness (complaints of hoarseness only on asking); 2 = moderate hoarseness (complaints of hoarseness on his/her own); 3 = severe hoarseness (hoarseness associated with throat pain)
Postoperative hoarseness | 24 hours after end of operation
  4-point scale, 0 = no hoarseness; 1 = mild hoarseness (complaints of hoarseness only on asking); 2 = moderate hoarseness (complaints of hoarseness on his/her own); 3 = severe hoarseness (hoarseness associated with throat pain)

CONTACTS AND LOCATIONS:
Overall Officials: Hansol KIM, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No